CLINICAL TRIAL: NCT04171986
Title: Mecapegfilgrastim Prevents Prospective, One-arm, Single-center Study of Concurrent Hyperfractionated Chemoradiotherapy With Neutropenia and Radiation Esophagitis in Limited-stage Small Cell Lung Cance
Brief Title: Mecapegfilgrastim Prevents Neutropenia and Radiation Esophagitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E2019367
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; HHPG-19K
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Group (Experimental)
  Interventions: Drug: Mecapegfilgrastim

INTERVENTIONS:
Drug: Mecapegfilgrastim — Mecapegfilgrastim; 6 mg, d7, q3w, total 2 cycles.

SUMMARY:
Evaluation of the efficacy and safety of Mecapegfilgrastim for the prevention of neutropenia and radiation esophagitis after hyperfractionation in patients with limited-stage small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with limited small cell lung cancer diagnosed by histopathology;
* ECOG 0-1 points;
* Weight ≥ 45 kg;
* Age 18-75 years old;
* It is expected that at least 2 cycles of EP chemotherapy will be completed as planned; once thiophene penicillin is used, chemotherapy should not be re-dosed within 12 days.
* Bone marrow hematopoietic function is normal, no bleeding tendency (INR<1.5);
* Laboratory tests are subject to: (1) Blood routine examination: Hb≥90g/L; WBC≥4.0×109/ L; ANC≥2.0×109/L; PLT≥100×109/L. (2) Liver function, biochemical examination: ALT and AST≤1.5×ULN; TBIL≤1.5×ULN; Serum creatinine≤1.5×ULN.
* According to the researcher's judgment, the test plan can be observed;
* Volunteer to participate in this clinical trial, understand the research process and be able to sign informed consent in writing.

Exclusion Criteria:

* There are currently uncontrolled infections or systemic antibiotics within 72 hours of receiving chemotherapy;
* Any abnormal bone marrow hyperplasia and other hematopoietic dysfunction;
* Patients who have received bone marrow or hematopoietic stem cell transplantation within the past 3 months;
* Patients with previous malignant tumors that have not been cured or have brain metastases;
* Liver function tests Total bilirubin (TBIL), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) are >2.5 times the upper limit of normal; if due to liver metastasis, the above indicators are >5 times the upper limit of normal;
* Renal function test: serum creatinine (Cr) > 1.5 times the upper limit of normal;
* Those who are allergic to this product;
* suffering from mental or neurological disorders that cannot be matched;
* Female patients during pregnancy or lactation; women of childbearing age who refuse to receive contraception;
* The investigator believes that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2019-11-10 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of neutrophil radiation esophagitis begins with hyperfractionated chemoradiotherapy. | 6 weeks
Incidence of 3 and 4 degrees neutropenia within 6 weeks from the start of hyperfractionated radiotherapy | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China